CLINICAL TRIAL: NCT06640231
Title: The Effect of XP-Endo Finisher Activation of Bioceramic Sealer on Postoperative Pain in Mandibular First Molar With Symptomatic Irreversible Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Amira Ali Fahmy Heteba, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUE.REC(21)/7-2024
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-10

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioceramic sealer activation with XP Endo Finisher. (Active Comparator)
  Interventions: Other: sealer activation after cleaning and shaping with XP-Endo Finisher
- Bioceramic sealer without activation. (Active Comparator)
  Interventions: Other: negative control where canals are obturated directly without sealer activation

INTERVENTIONS:
Other: sealer activation after cleaning and shaping with XP-Endo Finisher — activation of sealer before the obturation of root canals
  Arms: Bioceramic sealer activation with XP Endo Finisher.
Other: negative control where canals are obturated directly without sealer activation — sealer after cleaning and shaping before the obturation without using activation method
  Arms: Bioceramic sealer without activation.

SUMMARY:
The aim of endodontic obturation is to make a complete sealing along the length of the root canal system to ensuring the peri radicular tissue healing and sustained health. Disadvantages of gutta-percha-based root filling materials is lack of adhesiveness to canal wall dentin. So, a sealer or cement has to be used with gutta-percha to achieve a fluid-tight seal and fill the space between the canal wall dentin and the obturating material.

Drawbacks of resin-based sealer are difficult preparation technique of deep root canal cavity which also limit dentin bonding, difficult to be removed from the canal in retreatment cases and its shrinkage during setting.

Bio-ceramic root canal sealers become popular in recent years because of their unique chemical and physical properties. These sealers are consisting of biocompatible materials that resemble the of tooth structure natural composition so bio-ceramic sealers are an ideal choice for root canal treatment. Bio-ceramic sealers are better than traditional sealers due to their multiple physical properties for example excellent sealing ability, dimensional stability, and low solubility. These properties ensure that the sealers achieve a tight seal, inhibiting bacterial leakage and decreasing the risk of reinfection. Diaroot Bioaggregate (DiaDent), a white nanoparticle-sized ceramic cement composed of calcium silicate, calcium hydroxide and hydroxyapatite and considered a modified version of MTA, with the advantage of being aluminium-free in composition, a fact that contributes to its greater biocompatibility with periradicular tissue.Root canal sealers activation may improve their penetration into dentinal tubules and improve sealability and antimicrobial effects.

Recently, a non-tapered nickel-titanium rotary instrument (XP-endo Finisher; FKG, La Chaux-de-Fonds, Switzerland) has been designed to increase the efficiency in root canal wall cleaning specifically with limited impact on dentine throughout the literature, XP efficacy in decreasing microorganisms, dissolving organic tissue from artificial cavities in combination with NaOCl and penetrating into the isthmus has been analyzed.

The aim of this study to evaluate the effect of XP-Endo Finisher activation of Bioceramic sealer on postoperative pain in mandibular first molar with symptomatic irreversible pulpitis.

This study consists of 30 patients divided into 2 group each group having 15 patients.

Intervention:

Bioceramic sealer activation with XP Endo Finisher.

Control group:

Bioceramic sealer without activation.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 40 years old.
* No sex predilection.
* Patients seeking root canal treatment.
* Systematically healthy patient (ASA I, II).
* Patient who can understand numerical rate scale and sign an informed consent.
* Mandibular first molar teeth with:

  * Preoperative sharp (moderate or severe) pain.
  * Vital response of pulp tissue to cold pulp tester (ethyl chloride spray).
  * Normal periapical radiographic appearance.

Exclusion Criteria:

* Patients with American association of anesthesiologists (ASA) classification other than ASA T& II.
* Patients who have already ingested preoperative medication, such as analgesics, non-steroidal or steroidal anti-inflammatory drugs, within 12 hours of the start of treatment.
* Patients with NSAIDs allergy.
* Patients having two or more adjacent teeth needing root canal therapy.
* Pregnant patients.
* Patients with bleeding disorder.
* Patients with long term corticosteroid use
* Teeth having;

  * Necrotic pulp.
  * History or presence of swelling or fistulous tract.
  * Acute / chronic periapical abscess.
  * Mobility more than grade 1.
  * Pocket depth more than 5mm.
  * No possible restorability.
  * Previous root canal treatment.
  * Periapical radiolucency.
  * External or internal resorption.
  * Vertical root fracture.
* TMJ problems, bruxism, clenching or traumatic occlusion.
* Inability to understand and perform the given instructions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain after sealer activation with XP-Endo Finisher in comparison to without sealer activation | Immediately after obturation, 6-, 12-, 24- and 48-hours post-operative.
  Measuring of post-operative pain by Numerical rate scale(NRS) and pain level will be assigned to one of 4 categorical scores: None (0); Mild (1-3); Moderate (4-6); Severe (7-10).

SECONDARY OUTCOMES:
Number of analgesic tablets taken after endodontic treatment with sealer activation in comparison to without sealer activation | Up to 48 hours postoperatively.
  Measuring of number of analgesic tablets taken after endodontic treatment by counting.

OTHER OUTCOMES:
Lateral or periapical extrusion of sealer. | Immediately after obturation.
  detecting of lateral or periapical extrusion of sealer postoperative periapical radiograph.

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided